CLINICAL TRIAL: NCT04721561
Title: Robotic Assessment of Upper Limb Passive and Active Sensory Processing in the Chronic Phase After Stroke
Brief Title: Towards Understanding Upper Limb Rehabilitation After Stroke
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Prof. Dr., KU Leuven
Other Study IDs: S61997; C22/18/008 (Other Grant/Funding Number: KU Leuven C2 internal fund)
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Somatosensation; Sensory processing; Robotic assessment; Kinematics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic stroke patients: Patients who are at least 6 months after a first unilateral stroke
- Healthy controls: Healthy subjects with no history of any neurological condition and who are in the same age group as the chronic stroke patients

SUMMARY:
After a stroke, more than two out of three patients experience problems with upper limb movement and sensation. During the past decade, robotic technology has been increasingly used to asses these problems in a detailed and accurate manner. However, sensory processing, one of the most important sensory functions, has not been assessed using robotic technology yet. Therefore, the investigators have developed a robotic assessment of sensory processing. During this study, the investigators aim to initially validate this novel assessment. The investigators aim to examine 20 chronic stroke patients and 20 age-matched healthy controls using the robotic assessment on one hand, and a set of existing clinical assessments on the other hand. The investigators hypothesize that stroke patients will have a poorer performance on this novel robotic assessment compared to age-matched healthy controls, and that these findings are similar to what is found with existing clinical assessments.

DETAILED DESCRIPTION:
Up to 70% of stroke survivors show upper limb impairments consisting of motor and/or somatosensory impairments. These impairments often persist well into the chronic stage, and may lead to significant limitations in activities of daily living and may negatively affect quality of life. It is therefore of utmost importance to accurately assess upper limb impairments. Clinical assessments exist for both motor and somatosensory function, but lack good psychometric properties. Robotic technology show promising potential and is readily available to assess motor function and proprioception. Robotic assessment for sensory processing is currently not yet available, despite being the most relevant somatosensory function. Indeed, sensory processing shows the strongest association with upper limb movement, and only shows incomplete recovery at 6 months after stroke.

The investigators recently developed a novel robotic assessment of sensory processing, using the Kinarm End-Point Lab (BKIN Technologies Ltd., Canada). This cross-sectional study was set up to initially validate this novel robotic assessment and to collect pilot data to form the basis for future research. 20 chronic stroke patients and 20 age-matched controls will be recruited and will undergo extensive clinical and robotic assessment of upper limb motor and somatosensory function. The investigators hypothesize stoke patients with sensory processing deficits to have a worse performance on this novel robotic assessment compared to healthy controls and patients without sensory processing deficits. The investigators also hypothesize to see moderate to high correlations between the robotic assessment of sensory processing, and clinical assessments for both somatosensory and motor function.

ELIGIBILITY:
Inclusion Criteria - Stroke Patients:

* At least 18 years old
* A first-ever unilateral, supratentorial stroke (as defined by WHO)
* In the chronic phase after stroke (i.e. being at least 6 months after stroke)
* The ability to perform, at least to some extent, active shoulder abduction and wrist extension against gravity

Exclusion Criteria - Stroke Patients:

* Any serious musculoskeletal and/or other neurological conditions
* Serious communication or cognitive deficits
* No written informed consent

Inclusion Criteria - Healthy Controls:

- At least 18 years old

Exclusion Criteria - Healthy Controls:

* History of stroke or TIA
* Upper limb somatosensory and/or motor impairments
* Any serious musculoskeletal and/or other neurological conditions
* Serious communication or cognitive deficits
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from the community sample.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Kinarm: sensory processing task | Once in the chronic phase (at least 6 months after stroke)
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing

SECONDARY OUTCOMES:
Kinarm: position matching task | Once in the chronic phase (at least 6 months after stroke)
  Assessment of limb position sense using a 9-target mirror-matching task on the Kinarm End-Point Lab
Kinarm: visually guided reaching | Once in the chronic phase (at least 6 months after stroke)
  Assessment of motor function using a 4-target centre-out reaching task on the Kinarm End-Point Lab
Erasmus modified Nottingham sensory assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Tactile discrimination test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Tactile functional object recognition | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 42, with higher scores meaning better performance
Stereognosis section of the original Nottingham sensory assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 22, with higher scores meaning better performance
Wrist position sense test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of wrist position sense on a continuous scale, with lower scores meaning better performance
Perceptual threshold of touch | Once in the chronic phase (at least 6 months after stroke)
  TENS-based assessment of exteroception on a continuous scale, with lower scores meaning better performance
Fugl-Meyer upper extremity assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of motor function on an ordinal scale ranging from 0 to 66, with higher scores meaning better performance
Action research arm test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of motor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Barthel index | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of activities of daily living on an ordinal scale ranging from 0 to 20, with higher scores meaning better performance
Montreal cognitive assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of cognitive function on an ordinal scale ranging from 0 to 30, with higher scores meaning better performance
Star cancellation test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of visuospatial neglect on an ordinal scale ranging from 0 to 54, with higher scores meaning better performance, and a score below 44 indicating the presence of visuospatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided